CLINICAL TRIAL: NCT05929430
Title: Effects of a Mindfulness Program on the Occupational Balance and Mental Health of University Students. Protocol for a Randomized Controlled Trial Study. ATENEU Program (Mindfulness in University Students)
Brief Title: Mindfulness in University Students. ATENEU Program
Acronym: ATENEU
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Miguel Hernandez de Elche (Other)
Collaborators: Universidad Complutense de Madrid (Other)
Responsible Party: Principal Investigator, ALICIA SANCHEZ PEREZ, Associate Professor of Occupational Therapy, Universidad Miguel Hernandez de Elche
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: Mind02UMH
Record Dates: First submitted 2023-05-26; First posted 2023-07-03 (Actual); Last update posted 2024-12-24 (Actual); Status verified 2024-12

CONDITIONS: Occupational Balance; Mental Health Wellness; University Students; Burnout, Student
Keywords: Mindfulness; Occupational Balance; Mental Health; University Students; Burnout Student
MeSH Terms: conditions — Burnout, Psychological; Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: A randomized controlled clinical trial (RCT) with three arms
Who Masked: Care Provider, Investigator, Outcomes Assessor
Masking Description: Members of the research team who are not involved in the assessments and implementation of the intervention will be responsible for the random sequence and data analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Mindfulness-Based Health Care Program (MBHC). (Experimental): Mindfulness skills will take over a 6-week period. Mindfulness skills will deliver in a weekly group format. Participants will be instructed to follow mindfulness practice at home. The program is focused on cultivating mindfulness of present-moment, cultivating a nonreactive, nonjudgmental attitude toward the experience, and includes specific formal and informal practices aimed at cultivating healthy habits and lifestyle (e.g., activities of daily living such as feeding, bathing, or showering and other occupations such as communication management, health management, etc.; and prosocial components (e.g., kindness and compassion).
  Interventions: Behavioral: Mindfulness program
- Mindfulness-Based Health Care program with virtual reality (MBHC-VR). (Experimental): This program combines mindfulness practice with immersion in a virtual environment. The content and objectives of MBHC-VR program are the same that MBHC, with the main difference being that all formal practices of each session will be performed using VR.
  Interventions: Behavioral: Mindfulness program with Virtual Reality
- Waiting list control group (WL). (No Intervention): Participants in the WL control group will not receive any intervention during the study. However, for ethical reasons, at the end of the 3-month follow-up assessment, participants of this WL control group will be invited to participate in the MBHC program free of charge.

INTERVENTIONS:
Behavioral: Mindfulness program — Six weeks mindfulness program. The program is explained in arm descriptions.
  Arms: Mindfulness-Based Health Care Program (MBHC).
Behavioral: Mindfulness program with Virtual Reality — Six weeks mindfulness program. The program is explained in arm descriptions.
  Arms: Mindfulness-Based Health Care program with virtual reality (MBHC-VR).

SUMMARY:
The study aims to examine the effects of a mindfulness-based intervention and a mindfulness-based intervention with virtual reality on occupational balance and on the reduction of psychological distress in university students (i.e. stress, anxiety and depression). The specific objectives will be to examine the effects of the intervention on other variables related to mental health, psychological functioning and occupations, and their maintenance at three months.

DETAILED DESCRIPTION:
The college student population is considered at high risk for developing mental health problems with the prevalence of depression being 34%, anxiety 32%, and sleep disorders 33% post-pandemic. This psychological distress affects students worldwide and is linked to poor academic performance and the presence of health risk behaviors such as substance use or suicide. Addressing student mental health is an urgent research priority. As such, a growing number of universities are offering interventions aimed at students, including MBI or mindfulness which is defined as the ability to pay attention to present moment experience with interest, curiosity, and acceptance MBI has been shown to have beneficial effects in students but the level of adherence to the program is low. One of the possible solutions could be the incorporation of virtual reality (VR) due to the high affinity of this population with new technologies and the increase in its frequency of use in neurorehabilitation and clinical psychology.

Objectives:

The study aims to examine the effects of a mindfulness-based intervention and a mindfulness-based intervention with virtual reality on occupational balance and on the reduction of psychological distress in university students (i.e. stress, anxiety and depression). The specific objectives will be to examine the effects of the intervention on other variables related to mental health, psychological functioning and occupations, and their maintenance at three months.

Methodology:

Single-blind, 3-arm randomized clinical trial (RCT): traditional MBI, MBI with VR, passive control group (waiting list), with 4 evaluation moments: pre-intervention, inter-session, post-intervention and follow-up. Participants will be undergraduate, master and doctoral students of the Miguel Hernández University of Elche, Alicante.

Intervention: Mindfulness-Based Intervention, Mindfulness-Based Intervention with virtual reality and Control group.

Variables and instruments:

This study will be carried out with mixed methodology. The quantitative part will be carried out by means of ad hoc questionnaires and measurement instruments adapted and validated in Spain, and by means of EMA (Ecological Momentary Assessment).

The qualitative part will be conducted through Focus Groups.

ELIGIBILITY:
Inclusion Criteria:

* being 18 years old or older
* being a degree, master or doctorate student at Miguel Hernández University
* speaking fluent Spanish
* signing the informed consent form
* having attended at least 4 of the 6 sessions (66% of the program)
* internet access from a computer or smartphone to complete the online assessments and formal practices during the program.

Exclusion Criteria:

* miss more than 2 out of 6 sessions (33% of the program)
* present a severe mental disorder in active phase diagnosed by a health professional (e.g., schizophrenia, bipolar disorder)
* are under the influence of alcohol or other drugs during sessions and/or assessments (determined by the program instructor)
* participate in another standardized meditation program during the study period
* withdrew before starting the intervention.
* Additionally, should any participants require psychological or psychiatric treatment during the study, they will be excluded and referred to specialized care services.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 174 (Estimated)
Dates: Start 2023-11-02 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Change in Occupational Balance | Baseline (1 day), inter-session (one time per day over 42 days, from 1 week until 6 week), immediately post-intervention (6 weeks) and follow-up (18 weeks).
  Occupational Balance Questionnaire (OBQ) is a brief 13-item tool scored on a 6-point Likert-type response scale, ranging from 0 (strongly disagree) to 5 (strongly agree), with a total score ranging from 0 to 65, where a higher score indicates greater occupational balance. A question from the Ecological Momentary Assessment questionnaire will also be used to evaluate this variable in the inter-session time frame.
Change in Anxiety, Depression and Stress | Baseline (1 day), inter-session (one time per day over 42 days, from 1 week until 6 week), immediately post-intervention (6 weeks) and follow-up (18 weeks).
  Anxiety, Depression and Stress Scale (DASS 21) consists of 21 items, 7 items for each subscale: DASS-D (depression), DASS-A (anxiety) and DASS-S (stress). Participants are asked to rate the degree to which this statement has happened to them in the past week on a scale from 0 (has not happened to me) to 3 (has happened to me a lot or most of the time). A question from the Ecological Momentary Assessment questionnaire will also be used to evaluate this variable in the inter-session time frame.
Change in Academic stress | Baseline (1 day), inter-session (one time per day over 42 days, from 1 week until 6 week), immediately post-intervention (6 weeks) and follow-up (18 weeks).
  SISCO Inventory which consists of 31 items distributed into: 1 filter item (yes-no), 1 item on a Likert-type scale from 1 (a little) to 5 (a lot), 8 items on a Likert-type scale from 1 (never) to 5 (always) that allow identifying stressful stimuli, 15 items on a Likert-type scale from 1 (never) to 5 (always) allowing to identify stressful stimuli divided into physical, psychological and behavioural reactions and 6 items on a Likert-type scale from 1 (never) to 5 (always) allowing to identify the frequency of use of coping strategies. A question from the Ecological Momentary Assessment questionnaire will also be used to evaluate this variable in the inter-session time frame.
Change in Burnout | Baseline (1 day), inter-session (one time per day over 42 days, from 1 week until 6 week), immediately post-intervention (6 weeks) and follow-up (18 weeks).
  Maslach Burnout Inventory-Student Survey Questionnaire (MBI-SS). The MBI-SS contains 15 items grouped into 3 subscales: Emotional Exhaustion (5 items), Cynicism (4 items), and Academic Efficacy (6 items). These items are scored on a scale from 0 (never/never) to 6 (always/every day). High scores on burnout and cynicism and low scores on academic efficacy are indicative of burnout. A question from the Ecological Momentary Assessment questionnaire will also be used to evaluate this variable in the inter-session time frame.

SECONDARY OUTCOMES:
Change in Emotional dysregulation | Baseline (1 day), immediately post-intervention (6 weeks) and follow-up (18 weeks).
  Difficulties in Emotional Regulation Scale (DERS) contains 28 items grouped into 5 subscales: Attention-Inattention, Clarity-Confusion, Acceptance-Rejection, Functioning-Interference, and Regulation-Discontrol. These items are scored on a Likert-type scale from 1 (almost never) to 5 (almost always). Higher scores indicate greater difficulties in emotion regulation.
Change in Psychological flexibility | Baseline (1 day), immediately post-intervention (6 weeks) and follow-up (18 weeks).
  Acceptance and Action Questionnaire II (AAQ-II) consists of 7 items to which participants respond on a 7-point Likert-type scale from 1 (never true) to 7 (always true). Scores range from 7 to 49. Higher scores indicate a tendency to act on the need to control or avoid aversive thoughts, memories, or feelings.
Change in Mindfulness | Baseline (1 day), inter-session (one time per day over 42 days, from 1 week until 6 week), immediately post-intervention (6 weeks) and follow-up (18 weeks).
  Five Facets of Mindfulness Questionnaire Short-Form (FFMQ-SF) contains 24 items that assess the five facets of mindfulness: observing, describing, acting with awareness, non-judgement of inner experience, and non-reactivity to inner experience. It is scored on a Likert-type scale from 1 (never or very rarely true) to 5 (very often or always true). Higher scores indicate a greater capacity for mindfulness. A question from the Ecological Momentary Assessment questionnaire will also be used to evaluate this variable in the inter-session time frame.
Change in Self-compassion | Baseline (1 day), inter-session (one time per day over 42 days, from 1 week until 6 week), immediately post-intervention (6 weeks) and follow-up (18 weeks).
  Self-Compassion Scale short form (SCS-SF) consists of 12 items assessing 6 factors: Self-Kindness, Self-Judgment, Common Humanity, Isolation, Mindfulness, and Over-identification. Each item can be rated on a Likert-type scale from 1 (almost never) to 5 (almost always). Higher scores indicate greater self-compassion. A question from the Ecological Momentary Assessment questionnaire will also be used to evaluate this variable in the inter-session time frame.
Change in Life Satisfaction | Baseline (1 day), immediately post-intervention (6 weeks) and follow-up (18 weeks).
  Satisfaction with Life Scale (SLS) is composed of 5 items with a 7-point Likert-type scale (from 1, strongly disagree; to 7, strongly agree). The score ranges from 5 to 35, with higher scores indicating greater satisfaction.
Change in Adherence to the Mediterranean Diet | Baseline (1 day), immediately post-intervention (6 weeks) and follow-up (18 weeks).
  Mediterranean Diet Adherence Test is a brief dietary assessment instrument consisting of a set of 14 short questions whose evaluation is intended to provide information on adherence to the Mediterranean Diet pattern. This questionnaire scores one point per question, with a score of <9 meaning low adherence and a score of >=9 meaning good adherence.
Change in Sleep | Baseline (1 day), immediately post-intervention (6 weeks) and follow-up (18 weeks).
  Insomnia Severity Index (ISI) is a 5-item self-report instrument that assesses the severity of the sleep problem, the degree of dissatisfaction and the impact on quality of life. Scores range from 0 (best score) to 28 (worst score).
Change in Physical Activity | Baseline (1 day), immediately post-intervention (6 weeks) and follow-up (18 weeks).
  International Physical Activity Questionnaire (IPAQ-SF) is a self-administered questionnaire consisting of 7 items that assesses the time spent being physically active in the last 7 days.
Change in Mental representations | Baseline (1 day), immediately post-intervention (6 weeks) and follow-up (18 weeks).
  Plymouth Sensory Imagery Questionnaire (Psi-Q) consists of 21 items measuring 7 sensory modalities: vision, sound, smell, taste, touch, bodily sensation and emotions. The questionnaire has a Likert-type scale between 1 (no imagery) and 7 (perfectly clear and as vivid as the actual experience).

CONTACTS AND LOCATIONS:
Overall Officials: Alicia Sánchez Pérez, Ph.D, Principal Investigator — Universidad Miguel Hernández- Facultad de Medicina
Locations (1):
- Alicia Sánchez Pérez, Sant Joan d'Alacant, Alicante, Spain

IPD SHARING:
Plan to Share IPD: No
Three members of the research group will be in charge of data collection under the supervision of the principal investigator of this research project. All digital data, including evaluation questionnaires and consent forms, will be stored as a data package on an encrypted hard drive, strictly following the data management guidelines of the Research Ethics And Integrity Committee from Miguel Hernández Univesity. Identifiable personal data will be stored separately from anonymous data to avoid identification of personal data during handling. The confidentiality of the participants will be protected following the ethical guidelines of the Research Ethics And Integrity Committee from Miguel Hernández Univesity.
  Once all phases of data collection have been completed, the data will be analyzed by 2 members of the group. Data will be available upon request to the corresponding author once the study is completed.

REFERENCES:
- [Background] Sheldon E, Simmonds-Buckley M, Bone C, Mascarenhas T, Chan N, Wincott M, Gleeson H, Sow K, Hind D, Barkham M. Prevalence and risk factors for mental health problems in university undergraduate students: A systematic review with meta-analysis. J Affect Disord. 2021 May 15;287:282-292. doi: 10.1016/j.jad.2021.03.054. Epub 2021 Mar 26. PMID 33812241
- [Background] Yusoff MS, Abdul Rahim AF, Yaacob MJ. Prevalence and Sources of Stress among Universiti Sains Malaysia Medical Students. Malays J Med Sci. 2010 Jan;17(1):30-7. PMID 22135523
- [Background] Modrego-Alarcon M, Lopez-Del-Hoyo Y, Garcia-Campayo J, Perez-Aranda A, Navarro-Gil M, Beltran-Ruiz M, Morillo H, Delgado-Suarez I, Olivan-Arevalo R, Montero-Marin J. Efficacy of a mindfulness-based programme with and without virtual reality support to reduce stress in university students: A randomized controlled trial. Behav Res Ther. 2021 Jul;142:103866. doi: 10.1016/j.brat.2021.103866. Epub 2021 Apr 26. PMID 33957506
- [Background] Dhas BN, Wagman P. Occupational balance from a clinical perspective. Scand J Occup Ther. 2022 Jul;29(5):373-379. doi: 10.1080/11038128.2020.1865450. Epub 2020 Dec 31. PMID 33382004
- [Background] Regehr C, Glancy D, Pitts A. Interventions to reduce stress in university students: a review and meta-analysis. J Affect Disord. 2013 May 15;148(1):1-11. doi: 10.1016/j.jad.2012.11.026. Epub 2012 Dec 13. PMID 23246209
- [Background] Levit-Binnun N, Arbel K, Dorjee D. The Mindfulness Map: A Practical Classification Framework of Mindfulness Practices, Associated Intentions, and Experiential Understandings. Front Psychol. 2021 Oct 12;12:727857. doi: 10.3389/fpsyg.2021.727857. eCollection 2021. PMID 34712178
- [Background] Shapiro SL, Carlson LE, Astin JA, Freedman B. Mechanisms of mindfulness. J Clin Psychol. 2006 Mar;62(3):373-86. doi: 10.1002/jclp.20237. PMID 16385481
- [Background] Dawson AF, Brown WW, Anderson J, Datta B, Donald JN, Hong K, Allan S, Mole TB, Jones PB, Galante J. Mindfulness-Based Interventions for University Students: A Systematic Review and Meta-Analysis of Randomised Controlled Trials. Appl Psychol Health Well Being. 2020 Jul;12(2):384-410. doi: 10.1111/aphw.12188. Epub 2019 Nov 19. PMID 31743957
- [Background] Sanchez-Perez A, Mendialdua-Canales D, Hurtado-Pomares M, Peral-Gomez P, Juarez-Leal I, Espinosa-Sempere C, Fernandez-Pires P, Zango-Martin I, Abellan-Miralles I, Lopez-Gonzalez P, Valera-Gran D, Navarrete-Munoz EM. The ATENcion Plena en Enfermedad de Alzheimer (ATENEA-Mindfulness in Alzheimer's Disease) Program for Caregivers: Study Protocol for a Randomized Controlled Trial. Healthcare (Basel). 2022 Mar 15;10(3):542. doi: 10.3390/healthcare10030542. PMID 35327020
- [Derived] Lillo-Navarro C, Fernandez-Pires P, Benavides Gil G, Martinez-Zaragoza F, Chaves C, Roca P, Peral-Gomez P, Gonzalez Valero ME, Mendialdua Canales D, Poveda Alfaro JL, Goldin PR, Sanchez-Perez A. Effects of a mindfulness-based program on the occupational balance and mental health of university students. Protocol for a randomized controlled trial. PLoS One. 2024 May 2;19(5):e0302018. doi: 10.1371/journal.pone.0302018. eCollection 2024. PMID 38696406